CLINICAL TRIAL: NCT00870103
Title: An Evaluation of the Prophylactic Efficacy and Safety of the Administration of the Combination Formulation of Moxifloxacin 0.5% and Dexamethasone 0.1% Eye Drops in Inflammation and Infection Post-cataract Surgery
Brief Title: Study of Efficacy and Safety of Vigadexa in Treating Inflammation and Infection Post-cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Benny Li, Regional Scientific Clinical Affair Manager, Alcon Research Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-08-05
Record Dates: First submitted 2008-09-26; First posted 2009-03-26 (Estimated); Results first posted 2010-02-15 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Cataract
Keywords: Cataract
MeSH Terms: conditions — Cataract | interventions — Moxifloxacin; Dexamethasone; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vigadexa eye drops (Experimental): Vigadexa (moxifloxacin 0.5% and dexamethasone 0.1%) eye drops
  Interventions: Drug: Vigadexa (moxifloxacin 0.5% and dexamethasone 0.1%) eye drops

INTERVENTIONS:
Drug: Vigadexa (moxifloxacin 0.5% and dexamethasone 0.1%) eye drops — 1 drop every 6 hours into the study eye

SUMMARY:
To demonstrate that the combination formulation of Moxifloxacin/Dexamethasone Eye Drop is effective and safe for the prevention of postoperative inflammation as a consequence of cataract extraction surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≧18 years of age
* able to sign an informed consent and complete all required visits
* intends to have a cataract extraction surgery followed by implantation of a posterior chamber Intraocular lens (IOL)
* Intraocular Pressure (IOP) ≦ 20 millimeters mercury (mmHg)

Exclusion Criteria:

* Uncontrolled glaucoma or IOP
* use of ocular anti-infectious during the study and within 30 days prior to the enrollment, secondary implantation or replacement of IOL in the study eye
* use of steroid during the study or within 14 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 64 patients were enrolled into the study
Pre-assignment Details: Nonrandomized
Groups:
- Vigadexa Group: Vigadexa (moxifloxacin 0.5% and dexamethasone 0.1%) eye drops; 1 drop every 6 hours into the study eye
Period: Overall Study
Arm/Group | Vigadexa Group
Started | 64
Completed | 60
Not Completed | 4
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Vigadexa Group
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With a Score of Zero for Anterior Chamber Cells.
Description: The percentage of patients with a score of zero for Anterior chamber cells.
  Anterior chamber inflammation was evaluated based on the number of cells per high-power field measured using the narrowest slit beam of the lamp (0.5 at a height of 8mm).
  Anterior chamber cells was recorded on a 0-4 point scale,0 = Less than 5 cells; 1 = Mild: 5-10 cells; 2 = Moderate:11-20 cells; 3 = Marked: 21-50 cells; 4 = Severe: Greater than 50 cells / hypopyon
Time Frame: Day 15 after cataract surgery
Measure: Number; unit: Percentage of participants
Arm/Group | Vigadexa Group
Number analyzed (Participants) | 60
Percentage of participants | 91.7

2. Primary Outcome: The Percentage of Patients With no Ocular Pain
Time Frame: Day 15 after cataract surgery
Measure: Number; unit: Percentage of participants
Arm/Group | Vigadexa Group
Number analyzed (Participants) | 60
Percentage of participants | 96.7

ADVERSE EVENTS:
Arm/Group | Vigadexa Group
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No